CLINICAL TRIAL: NCT04645745
Title: Effects of Myo-inositol, Alpha-Lactalbumin and Folic Acid Treatment in PCOS Women of Mexico and Italy
Brief Title: Myo-inositol, Alpha-Lactalbumin and Folic Acid Treatment in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Collaborators: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Unfer Vittorio, Director, AGUNCO Obstetrics and Gynecology Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVittorio
Record Dates: First submitted 2020-07-23; First posted 2020-11-27 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Myo-inositol; alpha-lactalbumin; HOMA-index; ovulation; hyperandrogenism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Inositol; Lactalbumin; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- myo-inositol plus alpha-lactalbumin (Experimental): Patients were treated with 2 g myo-inositol, 50 mg alpha-LA and 200 mcg of Folic Acid twice a day for 6 months. Controls were the same patients at baseline (t0)
  Interventions: Dietary Supplement: myo-inositol, alpha-lactalbumin, folic acid

INTERVENTIONS:
Dietary Supplement: myo-inositol, alpha-lactalbumin, folic acid — Evaluating the improvement vs the baseline after three and six months of treatment

SUMMARY:
The main aim of this study is to evaluate the effect of myo-inositol and alpha-lactalbumin treatment on HOMA-index improvement in two different groups of women, belonging to the Mexican and Italian population, both affected by Polycystic Ovary Syndrome.

DETAILED DESCRIPTION:
This is an open-label clinical trial aimed at evaluating and comparing the effect of myo-inositol and alpha-lactalbumin treatment on HOMA-index improvement in two different groups of PCOS patients from the Mexican and Italian population. The addition of alpha-lactalbumin helps to increase the intestinal absorption of myo-inositol and consequently improve its effect. The scientific evidence so far available shows that these two groups of PCOS women have a different genetic, nutritional, and behavioural profile. Important factors are body mass index and insulin resistance, both increased in the Mexican women, although among them PCOS prevalence is not higher compared to many other populations. Therefore, the focus of this study is to check the effects of the combined administration of myo-inositol and alpha-lactalbumin for six months (with a control at three months) e to compare these effects between the two groups of patients, monitoring several hormonal parameters connected to the menstrual cycle regularization.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnosis based on the Rotterdam ESHRE-ASRM consensus workshop group1.
* Presence of Insulin resistance diagnosed by HOMA-Index
* Patients belonging to the Mexican population
* Patients belonging to the Italian population

Exclusion Criteria:

* BMI ≥ 30
* Other conditions causing ovulatory disorders and/or androgens hyper production such as: hyperprolactinemia, hypothyroidism, adrenal hyperplasia and Cushing syndrome
* Hormonal and/or pharmacological treatments in the previous 3 months that could interfere with ovulation
* Drastic changes in diet and physical activity
* Treatment with products containing inositols in the previous 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of Myo-inositol and alpha-lactalbumin treatment on HOMA-index | three and six months
  monitoring glucose and insulin levels in blood

SECONDARY OUTCOMES:
Evaluation of Myo-inositol and alpha-lactalbumin treatment on ovulation | three and six months
  dosage of Progesterone, LH, FSH.
Evaluation of Myo-inositol and alpha-lactalbumin treatment on hyperandrogenism | three and six months
  dosage of Total Testosterone, Free Testosterone, Androstenedione.

CONTACTS AND LOCATIONS:
Locations (2):
- AGUNCO Centre, Rome, Italy
- Hospital Juarez de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No